CLINICAL TRIAL: NCT02582242
Title: A 24-week, Multinational, Multicentre, Randomised, Open Label, Parallel-group Treat-to-target Trial to Compare Efficacy and Safety of Thrice Daily Versus Twice Daily NovoMix® 30 (Biphasic Insulin Aspart 30) in Subjects With Type 2 Diabetes Inadequately Controlled With Basal Insulin
Brief Title: Comparing Efficacy and Safety of Thrice Daily Versus Twice Daily NovoMix® 30 (Biphasic Insulin Aspart 30) in Subjects With Type 2 Diabetes Inadequately Controlled With Basal Insulin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-4200; U1111-1162-5508 (Other: WHO)
Record Dates: First submitted 2015-10-16; First posted 2015-10-21 (Estimated); Results first posted 2018-05-29 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: Diabetes; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BIAsp 30 TID (Experimental)
  Interventions: Drug: biphasic insulin aspart 30
- BIAsp 30 BID (Active Comparator)
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Administered subcutaneously (s.c., under the skin) thrice daily or twice daily. Subjects will continue with metformin all throughout the trial.

SUMMARY:
This trial is conducted in Asia. The aim of the trial is to compare efficacy and safety of thrice daily versus twice daily NovoMix® 30 (Biphasic insulin aspart 30) in subjects with type 2 diabetes inadequately controlled with basal insulin.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age at least 18 years at the time of signing informed consent. For Algeria only: age at least 19 years at the time of signing informed consent
* Type 2 diabetes subjects clinically diagnosed for at least 12 months prior to the day of screening (Visit 1)
* Treated with basal insulin for at least 90 days prior to the day of screening (Visit 1). The following basal insulin are allowed : insulin analogue once daily (OD) Neutral Protamine Hagedorn (NPH) OD or BID (twice daily)
* Treatment with metformin with or without one additional OAD (oral antidiabetic drug) for at least 90 days prior to the day of screening (Visit 1) Metformin must be at a stable dose of at least 1500 mg daily or maximum tolerated dose for at least 60 days prior to screening (Visit 1) One additional OAD:Sulphonylurea/Glinides/ a-glucosidase inhibitors/Dipeptidyl-peptidase-4 inhibitors/Sodium glucose co-transporter 2 (SGLT2) inhibitors (if applicable)
* HbA1c (glycosylated haemoglobin) 7.5%-10.0% (both inclusive) by central laboratory analysis at screening (Visit 1)
* Able and willing to intake three main meals daily (breakfast, lunch and main evening meal) throughout the trial. Definition of main meal as judged by the investigator

Exclusion Criteria:

* Previous insulin intensification regimen for more than 14 days: premixed insulin thrice daily, basal-bolus regimen or continuous subcutaneous insulin infusion (CSII). Treatment during hospitalisation or during gestational diabetes is allowed for periods longer than 14 days
* Anticipated initiation or change in concomitant medications for more than 14 consecutive days or on a frequent basis known to affect weight or glucose metabolism (e.g. orlistat, thyroid hormones, systemic corticosteroids)
* Impaired liver function, defined as alanine aminotransferase (ALT) equal to or above 2.5 times upper normal limit at screening (Visit 1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2017-03-18 (Actual); Study Completion 2017-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (39):
- Algeria (2):
  - Novo Nordisk Investigational Site, Algiers
  - Novo Nordisk Investigational Site, Oran
- China (18):
  - Novo Nordisk Investigational Site, Hefei, Anhui
  - Novo Nordisk Investigational Site, Beijing, Beijing Municipality
  - Novo Nordisk Investigational Site, Chongqing, Chongqing Municipality
  - Novo Nordisk Investigational Site, Fuzhou, Fujian
  - Novo Nordisk Investigational Site, Guangzhou, Guangdong
  - Novo Nordisk Investigational Site, Shenzhen, Guangdong
  - Novo Nordisk Investigational Site, Shijiazhuang, Hebei
  - Novo Nordisk Investigational Site, Changzhou, Jiangsu
  - Novo Nordisk Investigational Site, Nanjing, Jiangsu
  - Novo Nordisk Investigational Site, Suzhou, Jiangsu
  - Novo Nordisk Investigational Site, Wuxi, Jiangsu
  - Novo Nordisk Investigational Site, Zhenjiang, Jiangsu
  - Novo Nordisk Investigational Site, Nanchang, Jiangxi
  - Novo Nordisk Investigational Site, Changchun, Jilin
  - Novo Nordisk Investigational Site, Dalian, Liaoning
  - Novo Nordisk Investigational Site, Shanghai, Shanghai Municipality
  - Novo Nordisk Investigational Site, Chengdu, Sichuan
  - Novo Nordisk Investigational Site, Tianjin, Tianjin Municipality
- Novo Nordisk Investigational Site, Shatin, New Territories, Hong Kong
- India (7):
  - Novo Nordisk Investigational Site, Visakhapatnam, Andhra Pradesh
  - Novo Nordisk Investigational Site, Guwahati, Assam
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Mysore, Karnataka
  - Novo Nordisk Investigational Site, Madurai, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, New Delhi
- Taiwan (3):
  - Novo Nordisk Investigational Site, Kaohsiung City
  - Novo Nordisk Investigational Site, Taichung
  - Novo Nordisk Investigational Site, Taipei
- Turkey (Türkiye) (4):
  - Novo Nordisk Investigational Site, Adana
  - Novo Nordisk Investigational Site, Bursa
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Kahramanmaraş
- Ukraine (4):
  - Novo Nordisk Investigational Site, Dnipro
  - Novo Nordisk Investigational Site, Kiev
  - Novo Nordisk Investigational Site, Lviv
  - Novo Nordisk Investigational Site, Ternopil

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://www.novonordisk-trials.com/website/content/how-to-access-clinical-trial-datasets.aspx

REFERENCES:
- [Result] Yang W, Ersoy C, Wang G, Ye S, Liu J, Miao H, Asirvatham A, Werther S, Kadu P, Chow F. Efficacy and safety of three-times-daily versus twice-daily biphasic insulin aspart 30 in patients with type 2 diabetes mellitus inadequately controlled with basal insulin combined with oral antidiabetic drugs. Diabetes Res Clin Pract. 2019 Apr;150:158-166. doi: 10.1016/j.diabres.2019.02.023. Epub 2019 Mar 11. PMID 30872064
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 50 sites were approved for recruiting subjects, of which 48 sites (in 2 regions) screened and randomized the subjects (China region, including mainland China, Hong Kong and Taiwan; non-China region, including other 4 countries) as follows: Algeria: 3; mainland China: 23; Hong Kong: 1; India: 8; Taiwan: 4; Turkey: 5; Ukraine: 4.
Groups:
- Biphasic Insulin Aspart 30 (Three Times Daily): Subjects received biphasic insulin aspart 30 (BIAsp 30; a mixture of soluble insulin aspart [IAsp] 30% and protaminated IAsp 70%) three times daily (TID); before breakfast, lunch and main evening meal for a duration of 24-week. BIAsp 30 was administered as subcutaneous (s.c.; under the skin) injection according to the locally approved label and as described in the direction for use. The total daily dose of pre-trial basal insulin was transferred to the total daily starting dose of BIAsp 30 by unit-to-unit, which was distributed along meals at the investigator's discretion. During the 24-week treatment period, the insulin dose was individually titrated on a weekly basis for all subjects in order to achieve the pre-meal self-measured plasma glucose (SMPG) target of 4.4-6.1 mmol/L (80-110 mg/dL). Subjects continued with their stable, pre-trial dose of metformin (a total daily oral dose of >=1500 mg metformin or maximum tolerated dose) throughout the entire treatment period.
- Biphasic Insulin Aspart 30 (Twice Daily): Subjects received BIAsp 30 twice daily (BID); before breakfast and main evening meal for a duration of 24-week. BIAsp 30 was administered as s.c. injection according to the locally approved label and as described in the direction for use. The total daily dose of pre-trial basal insulin was transferred to the total daily starting dose of BIAsp 30 by unit-to-unit, which was distributed along meals at the investigator's discretion. During the 24-week treatment period, the insulin dose was individually titrated on a weekly basis for all subjects in order to achieve the pre-meal SMPG target of 4.4-6.1 mmol/L (80-110 mg/dL). Subjects continued with their stable, pre-trial dose of metformin (a total daily oral dose of >=1500 mg metformin or maximum tolerated dose) throughout the entire treatment period.
Period: Overall Study
Arm/Group | Biphasic Insulin Aspart 30 (Three Times Daily) | Biphasic Insulin Aspart 30 (Twice Daily)
Started | 220 | 217
Completed | 200 | 200
Not Completed | 20 | 17
Not completed — Adverse Event | 4 | 3
Not completed — Protocol Violation | 3 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 11 | 11
Not completed — Unclassified | 2 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomised subjects who were dosed and had any post randomisation data.
Groups:
- Biphasic Insulin Aspart 30 (Three Times Daily): Subjects received BIAsp 30 TID; before breakfast, lunch and main evening meal for a duration of 24-week. BIAsp 30 was administered as s.c. injection according to the locally approved label and as described in the direction for use. The total daily dose of pre-trial basal insulin was transferred to the total daily starting dose of BIAsp 30 by unit-to-unit, which was distributed along meals at the investigator's discretion. During the 24-week treatment period, the insulin dose was individually titrated on a weekly basis for all subjects in order to achieve the pre-meal SMPG target of 4.4-6.1 mmol/L (80-110 mg/dL). Subjects continued with their stable, pre-trial dose of metformin (a total daily oral dose of >=1500 mg metformin or maximum tolerated dose) throughout the entire treatment period.
- Biphasic Insulin Aspart 30 (Twice Daily): Subjects received BIAsp 30 BID; before breakfast and main evening meal for a duration of 24-week. BIAsp 30 was administered as s.c. injection according to the locally approved label and as described in the direction for use. The total daily dose of pre-trial basal insulin was transferred to the total daily starting dose of BIAsp 30 by unit-to-unit, which was distributed along meals at the investigator's discretion. During the 24-week treatment period, the insulin dose was individually titrated on a weekly basis for all subjects in order to achieve the pre-meal SMPG target of 4.4-6.1 mmol/L (80-110 mg/dL). Subjects continued with their stable, pre-trial dose of metformin (a total daily oral dose of >=1500 mg metformin or maximum tolerated dose) throughout the entire treatment period.
- Total: Total of all reporting groups
Arm/Group | Biphasic Insulin Aspart 30 (Three Times Daily) | Biphasic Insulin Aspart 30 (Twice Daily) | Total
Number analyzed (Participants) | 220 | 217 | 437
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (9.8) | 56.6 (9.3) | 56.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 108 | 220
  Male | 108 | 109 | 217
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 218 | 217 | 435
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 181 | 170 | 351
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 39 | 47 | 86
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] | 8.74 (0.69) | 8.68 (0.69) | 8.71 (0.69)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 8.68 (2.68) | 8.72 (2.39) | 8.70 (2.54)
Body weight [Mean (Standard Deviation); unit: kg] | 71.57 (13.38) | 72.24 (13.01) | 71.90 (13.19)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Description: Change from baseline in HbA1c was evaluated after 24 weeks of treatment. Missing data was imputed using the last observation carried forward (LOCF) method.
Time Frame: Week 0, Week 24
Population: FAS included all randomised subjects who were dosed and had any post randomisation data.
Measure: Mean (Standard Deviation); unit: Percentage (%) of HbA1c
Arm/Group | Biphasic Insulin Aspart 30 (Three Times Daily) | Biphasic Insulin Aspart 30 (Twice Daily)
Number analyzed (Participants) | 220 | 217
Percentage (%) of HbA1c | -1.66 (1.00) | -1.52 (0.94)
Statistical Analysis 1: Comparison: Biphasic Insulin Aspart 30 (Three Times Daily) vs Biphasic Insulin Aspart 30 (Twice Daily); The analysis was based on a mixed-effect model for repeated measures including changes from baseline in HbA1c at visit 6, 10, 14, 18, 22 and 26 (in week 4, 8, 12, 16, 20 and 24, respectively). The model included treatment, strata and region as fixed factors, subject as random effect, baseline HbA1c as covariate and interaction between all fixed effects and visit, and between the covariate and visit; Test type: Other; p = 0.2601, Mixed model for repeated measurements; Treatment difference at week 24 = -0.09, 95% CI 2-sided [-0.23 to 0.06] — Treatment difference at week 24: BIAsp 30 (TID) - BIAsp 30 (BID). Number of subjects contributed to the statistical analysis: N=217 for BIAsp 30 (TID) and N=213 for BIAsp 30 (BID)

2. Secondary Outcome: Proportion of Subjects Achieving HbA1c Below 7.0%
Description: Percentage of subjects achieving HbA1c <7.0% (yes or no) was evaluated after 24 weeks of treatment.
Time Frame: Week 24
Population: FAS included all randomised subjects who were dosed and had any post randomisation data.
Measure: Number; unit: Percentage (%) of participants
Arm/Group | Biphasic Insulin Aspart 30 (Three Times Daily) | Biphasic Insulin Aspart 30 (Twice Daily)
Number analyzed (Participants) | 220 | 217
Percentage (%) of participants
  Yes | 54.5 | 47.5
  No | 45.5 | 52.5

3. Secondary Outcome: Proportion of Subjects Achieving HbA1c Below 7.0% Without Severe Hypoglycaemic Episodes.
Description: Percentage of subjects achieving HbA1c <7.0% (yes or no) without severe hypoglycaemic episodes was evaluated after 24 weeks of treatment. Severe hypoglycaemia: Episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. Plasma glucose (PG) concentrations may not be available during event, but neurological recovery following return of PG to normal is considered sufficient evidence that the event was induced by low PG concentration.
Time Frame: Week 24
Population: FAS included all randomised subjects who were dosed and had any post randomisation data.
Measure: Number; unit: Percentage (%) of participants
Arm/Group | Biphasic Insulin Aspart 30 (Three Times Daily) | Biphasic Insulin Aspart 30 (Twice Daily)
Number analyzed (Participants) | 220 | 217
Percentage (%) of participants
  Yes | 50.0 | 44.7
  No | 50.0 | 55.3

4. Secondary Outcome: Proportion of Subjects Achieving HbA1c Below 7.0% Without Severe or Blood Glucose (BG) Confirmed Hypoglycaemic Episodes (According to the Novo Nordisk Classification)
Description: Percentage of subjects achieving HbA1c <7.0% (yes or no) without severe or BG confirmed hypoglycaemic episodes (according to the Novo Nordisk classification) was evaluated after 24 weeks of treatment. Severe or BG confirmed hypoglycaemia: an episode that is severe according to the American Diabetes Association (ADA) classification or BG confirmed by a plasma glucose (PG) value <3.1 mmol/L (56 mg/dL) with or without symptoms consistent with hypoglycaemia. Severe hypoglycaemia as per ADA: Episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. PG concentrations may not be available during event, but neurological recovery following return of PG to normal is considered sufficient evidence that the event was induced by low PG concentration.
Time Frame: Week 24
Population: FAS included all randomised subjects who were dosed and had any post randomisation data.
Measure: Number; unit: Percentage (%) of participants
Arm/Group | Biphasic Insulin Aspart 30 (Three Times Daily) | Biphasic Insulin Aspart 30 (Twice Daily)
Number analyzed (Participants) | 220 | 217
Percentage (%) of participants
  Yes | 27.3 | 21.7
  No | 72.7 | 78.3

5. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes Classified According to the American Diabetes Association (ADA) Definition
Description: ADA classification of hypoglycaemia:
  1. Severe:Episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. PG concentrations may not be available during event, but neurological recovery following return of PG to normal is considered sufficient evidence that the event was induced by low PG concentration
  2. Asymptomatic:Episode not accompanied by typical symptoms of hypoglycaemia, but with a measured PG concentration ≤3.9 mmol/L
  3. Documented symptomatic:Episode during which typical symptoms of hypoglycaemia are accompanied by a measured PG concentration ≤3.9 mmol/L
  4. Pseudo:Episode during which person with diabetes reports any of the typical symptoms of hypoglycaemia with measured PG concentration >3.9 mmol/L but approaching that level
  5. Probable symptomatic:Episode during which symptoms of hypoglycaemia are not accompanied by PG determination but that was presumably caused by a PG concentration ≤3.9 mmol/L
Time Frame: Week 0-24
Population: Safety analysis set included all subjects who received at least one dose of investigational product (BIAsp 30). Treatment emergent hypoglycaemic episodes were defined as the hypoglycaemic episodes, which occurred on or after the first day of trial product administration (in week 0), and no later than 7 days after the last day on trial product.
Measure: Number; unit: Count of hypoglycaemic episodes
Arm/Group | Biphasic Insulin Aspart 30 (Three Times Daily) | Biphasic Insulin Aspart 30 (Twice Daily)
Number analyzed (Participants) | 220 | 217
Count of hypoglycaemic episodes
  Severe | 3 | 3
  Asymptomatic | 397 | 344
  Documented symptomatic | 642 | 765
  Pseudo-hypoglycaemia | 54 | 93
  Probable symptomatic | 61 | 30

6. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes Classified According to Novo Nordisk Definition
Description: Treatment emergent hypoglycaemic episodes were defined as the hypoglycaemic episodes, which occurred on or after the first day of trial product administration (in week 0), and no later than 7 days after the last day on trial product.
  Novo Nordisk (NN) classification of hypoglycaemia:
  1. Severe hypoglycaemia: According to the ADA classification.
  2. Blood glucose (BG) confirmed hypoglycaemia: an episode that is BG confirmed by a plasma glucose value <3.1 mmol/L (56 mg/dL) with or without symptoms consistent with hypoglycaemia.
  3. Severe or BG confirmed hypoglycaemia: an episode that is severe according to the ADA classification or BG confirmed by a plasma glucose value <3.1 mmol/L (56 mg/dL) with or without symptoms consistent with hypoglycaemia.
Time Frame: Week 0-24
Population: Safety analysis set included all subjects who received at least one dose of investigational product (BIAsp 30).
Measure: Number; unit: Count of hypoglycaemic episodes
Arm/Group | Biphasic Insulin Aspart 30 (Three Times Daily) | Biphasic Insulin Aspart 30 (Twice Daily)
Number analyzed (Participants) | 220 | 217
Count of hypoglycaemic episodes
  Severe | 3 | 3
  BG confirmed | 249 | 249
  Severe or BG confirmed | 252 | 252
  Severe or BG confirmed symptomatic | 195 | 223
  NN unclassifiable | 905 | 983

7. Secondary Outcome: Change From Baseline in FPG by Central Laboratory Analysis
Description: Change from baseline in fasting plasma glucose (FPG) by central laboratory analysis was evaluated after 24 weeks of treatment. Missing data was imputed using the LOCF method.
Time Frame: Week 0, Week 24
Population: FAS included all randomised subjects who were dosed and had any post randomisation data. Number analyzed = number of subjects contributed to the evaluation at the specified time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Biphasic Insulin Aspart 30 (Three Times Daily) | Biphasic Insulin Aspart 30 (Twice Daily)
Number analyzed (Participants) | 220 | 217
mmol/L | -1.34 (3.10) | -1.07 (2.64)

8. Secondary Outcome: 7-point SMPG Profile
Description: 7-point self-measured plasma glucose (SMPG) profiles was evaluated after 24 weeks of treatment.
  Subjects were instructed to perform the following SMPG measurements:
  1. Before breakfast.
  2. 120 minutes after the start of breakfast.
  3. Before lunch.
  4. 120 minutes after the start of lunch.
  5. Before main evening meal.
  6. 120 minutes after the start of main evening meal.
  7. At bedtime. Missing data was imputed using the LOCF method.
Time Frame: Week 24
Population: FAS included all randomised subjects who were dosed and had any post randomisation data. Number analyzed = number of subjects contributed to the evaluation at specified time points.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Biphasic Insulin Aspart 30 (Three Times Daily) | Biphasic Insulin Aspart 30 (Twice Daily)
Number analyzed (Participants) | 220 | 217
mmol/L
  Before breakfast: number analyzed (Participants) | 219 | 212
  Before breakfast | 6.87 (1.61) | 6.86 (1.71)
  120 minutes after start of breakfast: number analyzed (Participants) | 215 | 208
  120 minutes after start of breakfast | 9.33 (3.14) | 9.04 (3.20)
  Before lunch: number analyzed (Participants) | 217 | 214
  Before lunch | 6.86 (2.21) | 7.09 (2.72)
  120 minutes after start of lunch: number analyzed (Participants) | 216 | 211
  120 minutes after start of lunch | 9.48 (3.02) | 9.92 (3.54)
  Before main evening meal: number analyzed (Participants) | 219 | 213
  Before main evening meal | 7.26 (2.08) | 7.68 (2.53)
  120 minutes after start of main evening meal: number analyzed (Participants) | 217 | 208
  120 minutes after start of main evening meal | 8.77 (3.00) | 9.09 (3.29)
  At bedtime: number analyzed (Participants) | 211 | 207
  At bedtime | 7.69 (2.50) | 8.24 (3.15)

9. Secondary Outcome: 7-point SMPG Profiles: Change From Baseline in 2-hour PPG at Individual Meal (Breakfast, Lunch and Main Evening Meal)
Description: Change from baseline in 2-hour postprandial glucose (PPG) at individual meal (breakfast, lunch and main evening meal) was evaluated after 24 weeks of treatment. Missing data was imputed using the LOCF method.
Time Frame: Week 0, Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Biphasic Insulin Aspart 30 (Three Times Daily) | Biphasic Insulin Aspart 30 (Twice Daily)
Number analyzed (Participants) | 220 | 217
mmol/L
  Change in PPG breakfast: number analyzed (Participants) | 215 | 208
  Change in PPG breakfast | -4.17 (4.84) | -4.03 (4.22)
  Change in PPG lunch: number analyzed (Participants) | 216 | 215
  Change in PPG lunch | -3.43 (4.56) | -3.27 (4.59)
  Change in PPG main evening meal: number analyzed (Participants) | 216 | 214
  Change in PPG main evening meal | -4.38 (4.44) | -4.09 (4.71)

10. Secondary Outcome: 7-point SMPG Profiles: Change From Baseline in PPG Increment at Individual Meal (Breakfast, Lunch and Main Evening Meal)
Description: Change from baseline in PPG increment at individual meal (breakfast, lunch and main evening meal) was evaluated after 24 weeks of treatment. Missing data was imputed using the LOCF method.
Time Frame: Week 0, Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Biphasic Insulin Aspart 30 (Three Times Daily) | Biphasic Insulin Aspart 30 (Twice Daily)
Number analyzed (Participants) | 220 | 217
mmol/L
  Change in PPG increment breakfast: number analyzed (Participants) | 215 | 207
  Change in PPG increment breakfast | -2.06 (4.44) | -2.02 (3.95)
  Change in PPG increment lunch: number analyzed (Participants) | 216 | 211
  Change in PPG increment lunch | -0.13 (4.38) | -0.14 (4.40)
  Change in PPG increment main evening meal: number analyzed (Participants) | 216 | 211
  Change in PPG increment main evening meal | -0.64 (4.55) | -1.60 (4.72)

11. Secondary Outcome: 7-point SMPG Profiles: Change From Baseline in Mean of 2-hour PPG Over 3 Main Meals (Breakfast, Lunch and Main Evening Meal)
Description: Change from baseline in mean of 2-hour PPG at individual meal (breakfast, lunch and main evening meal) was evaluated after 24 weeks of treatment. Missing data was imputed using the LOCF method.
Time Frame: Week 0, Week 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Biphasic Insulin Aspart 30 (Three Times Daily) | Biphasic Insulin Aspart 30 (Twice Daily)
Number analyzed (Participants) | 220 | 217
mmol/L | -3.98 (3.59) | -3.77 (3.48)

12. Secondary Outcome: 7-point SMPG Profiles: Change From Baseline in Mean of PPG Increment Over 3 Main Meals (Breakfast, Lunch and Main Evening Meal)
Description: Change from baseline in mean of PPG increment at individual meal (breakfast, lunch and main evening meal) was evaluated after 24 weeks of treatment. Missing data was imputed using the LOCF method.
Time Frame: Week 0, Week 24
Population: FAS included all randomised subjects who were dosed and had any post randomisation data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Biphasic Insulin Aspart 30 (Three Times Daily) | Biphasic Insulin Aspart 30 (Twice Daily)
Number analyzed (Participants) | 220 | 217
mmol/L | -0.96 (2.53) | -1.22 (2.68)

13. Secondary Outcome: 7-point SMPG Profiles: Change From Baseline in Mean of the 7-point Profile
Description: Change from baseline in mean of the 7-point SMPG profiles was evaluated after 24 weeks of treatment. Missing data was imputed using the LOCF method.
Time Frame: Week 0, Week 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Biphasic Insulin Aspart 30 (Three Times Daily) | Biphasic Insulin Aspart 30 (Twice Daily)
Number analyzed (Participants) | 220 | 217
mmol/L | -3.58 (3.08) | -3.27 (2.84)

14. Secondary Outcome: 7-point SMPG Profiles: Fluctuation in the 7-point Profile
Description: Fluctuation in the 7-point SMPG profile was evaluated after 24 weeks of treatment. Fluctuation in 7-point SMPG profile was the average absolute difference to the mean of the profile of the 7-point SMPG measurements accumulated over the profile. Missing data was imputed using the LOCF method.
Time Frame: Week 24
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mmol/L
Arm/Group | Biphasic Insulin Aspart 30 (Three Times Daily) | Biphasic Insulin Aspart 30 (Twice Daily)
Number analyzed (Participants) | 220 | 217
mmol/L | 1.04 (54.04) | 1.05 (54.39)

15. Secondary Outcome: Incidence of Treatment Emergent Adverse Events (TEAEs)
Description: Incidence of TEAEs was recorded during 24 weeks of treatment. A TEAE was defined as an event that has onset date (or increase in severity) on or after the first day of exposure to trial product (in week 0) and no later than 7 days after the last day on trial product.
Time Frame: Week 0-24
Population: Safety analysis set included all subjects who received at least one dose of investigational product (BIAsp 30). Number analyzed = number of subjects with corresponding numbers of TEAEs.
Measure: Number; unit: Number of adverse events
Arm/Group | Biphasic Insulin Aspart 30 (Three Times Daily) | Biphasic Insulin Aspart 30 (Twice Daily)
Number analyzed (Participants) | 220 | 217
Number of adverse events | 275 | 251

16. Secondary Outcome: Total Daily Insulin Dose
Description: Total daily insulin dose was the sum of doses given before breakfast and before main evening meal for the BID treatment group, and the sum of doses given before breakfast, before lunch and before main evening meal for the TID treatment group. Missing data was imputed using the LOCF method.
Time Frame: Week 1, Week 24
Population: Safety analysis set included all subjects who received at least one dose of investigational product (BIAsp 30). Number analyzed = number of subjects contributed to the evaluation at the specified time point.
Measure: Mean (Standard Deviation); unit: Units (U)
Arm/Group | Biphasic Insulin Aspart 30 (Three Times Daily) | Biphasic Insulin Aspart 30 (Twice Daily)
Number analyzed (Participants) | 220 | 217
Units (U)
  Week 1: number analyzed (Participants) | 220 | 216
  Week 1 | 24.5 (10.0) | 24.2 (13.0)
  Week 24 | 67.4 (35.5) | 63.4 (33.1)

17. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight was evaluated after 24 weeks of treatment. Missing data was imputed using the LOCF method.
Time Frame: Week 0, Week 24
Population: Safety analysis set included all subjects who received at least one dose of investigational product (BIAsp 30).
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Biphasic Insulin Aspart 30 (Three Times Daily) | Biphasic Insulin Aspart 30 (Twice Daily)
Number analyzed (Participants) | 220 | 217
Kilogram (kg) | 1.45 (3.11) | 1.65 (2.85)

18. Secondary Outcome: Change From Baseline in Patient-reported Treatment Satisfaction as Assessed by the Diabetes Treatment Satisfaction Questionnaire (Status) (DTSQs)
Description: Change from baseline in patient-reported treatment satisfaction (as assessed by the DTSQs) was evaluated after 24 weeks of treatment. The DTSQs is a self-completion questionnaire used to investigate the subject's treatment satisfaction. The DTSQ contained 8 questions, which were scored on a scale from 0 to 6. Out of 8 questions, 6 were related to the overall treatment satisfaction and 2 were related to glycaemic control (hypoglycaemia and hyperglycaemia). Results for the 6 questions relating to overall treatment satisfaction are presented together whereas the 2 questions relating to blood glucose are presented separately. For the overall treatment satisfaction, a higher score (0-36) was related to a better perception of treatment satisfaction. For hypoglycaemia and hyperglycaemia, a lower score (0-6) was related to a better blood glucose control. Missing data was imputed using the LOCF method.
Time Frame: Week 0, Week 24
Population: FAS included all randomised subjects who were dosed and had any post randomisation data.
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Biphasic Insulin Aspart 30 (Three Times Daily) | Biphasic Insulin Aspart 30 (Twice Daily)
Number analyzed (Participants) | 220 | 217
Score on a scale
  Overall treatment satisfaction | 2 [-29 to 24] | 4 [-21 to 29]
  Hypoglycaemia | 0 [-6 to 6] | 0 [-5 to 6]
  Hyperglycaemia | -1 [-6 to 4] | -1 [-6 to 5]

ADVERSE EVENTS:
Time Frame: Week 0 to week 24 + 7 days. All AEs are treatment emergent, i.e., TEAEs.
Description: Results are based on the safety analysis set, which included all subjects who received at least one dose of investigational product (BIAsp 30).
Arm/Group | Biphasic Insulin Aspart 30 (Three Times Daily) | Biphasic Insulin Aspart 30 (Twice Daily)
All-Cause Mortality (participants affected / at risk) | 0/220 | 0/217
Serious Adverse Events (participants affected / at risk) | 12/220 | 9/217
Other Adverse Events (participants affected / at risk) | 34/220 | 36/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biphasic Insulin Aspart 30 (Three Times Daily) (N=220) | Biphasic Insulin Aspart 30 (Twice Daily) (N=217)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1)
Hypoglycaemic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biphasic Insulin Aspart 30 (Three Times Daily) (N=220) | Biphasic Insulin Aspart 30 (Twice Daily) (N=217)
Headache (Nervous system disorders) | 10 (16) | 11 (13)
Upper respiratory tract infection (Infections and infestations) | 26 (31) | 27 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/42/NCT02582242/Prot_SAP_000.pdf